CLINICAL TRIAL: NCT06543511
Title: MyeloGen: Germline Testing for Predisposition to Myeloid Malignancies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Contractual issues. Will be re-submitted as new protocol.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Reilly, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-087
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Myeloid Malignancy; Myeloid Malignancies; Blood Cancer; Blood Cancers
Keywords: Myeloid Malignancy; Myeloid Malignancies; Blood Cancer; Blood Cancers
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Germline Genetic Testing (Experimental): Participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with educational video and questionnaires.
  * Skin punch biopsy.
  * Genetic testing results.
  * Surveys and questionnaires.
  * Follow up via medical records for up to 2 years from time of study consent.
  Interventions: Other: Genetic Blood Test

INTERVENTIONS:
Other: Genetic Blood Test — Germline genetic testing using skin fibroblasts
  Other Names: Custom Hereditary Cancer Gene Panel

SUMMARY:
This research study is evaluating the feasibility of conducting cancer genetic testing using healthy skin cells among participants with a diagnosis of a blood cancer. Additionally, investigators will evaluate how often participants with blood cancers are found to have risk for cancer based on family genes.

DETAILED DESCRIPTION:
The purpose of this prospective, non-randomized, non-therapeutic, single arm study is to determine the feasibility and benefit of performing genetic testing for all participants with a blood cancer diagnosis regardless of clinical suspicion.

Research study procedures include screening for eligibility, in-clinic visits, questionnaires, and skin punch biopsies. Participants will receive germline genetic testing with a comprehensive hereditary cancer gene panel.

It is expected that about 200 individuals with blood cancer will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Participants must have histologically confirmed myeloid malignancy OR bone marrow failure within the last 6 months prior to screening.
* Ability to understand and provide a signed and completed consent document in English or Spanish.

Exclusion Criteria:

* Patients with who cannot safely undergo skin biopsy as adjudicated by the study team.
* Patients who have previously undergone germline genetic testing for predisposition to myeloid malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-29 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Genetic Testing Completion Rate | Up to 63 months
  Feasibility is defined as a minimum of 75% of consented participants complete germline genetic testing with the return of test results within 10 weeks of study consent.
Incidence Rate of Positive Genetic Results | Up to 63 months
  Defined as the proportion of participants with a "positive" result on the germline genetic testing. Positive results equal Variants classified as Pathogenic (P), Likely pathogenic (LP), or Variants of Uncertain Significance (VUS) with supporting pathogenic criteria.

SECONDARY OUTCOMES:
Participant Knowledge of Genetic Testing Pre-Education | At baseline
  Assessed by the KnowGene6 questionnaire, a 6-question survey assessing participant understanding of inherited genetic risk. Responses will be summarized by question and the number of correct answers will be compared.
Participant Knowledge of Genetic Testing Post-Education | At baseline, following pre-educational video
  Assessed by the KnowGene6 questionnaire, a 6-question survey assessing participant understanding of inherited genetic risk. Responses will be summarized by question and the number of correct answers will be compared.
Participant Satisfaction Score on Genetic Testing Satisfaction (GTS) Survey 1 | At baseline
  Assessed by the Genetic Testing Satisfaction (GTS) 1, a 10-item measure rated on a 5-point scale from 1 "Strongly Disagree" to 5 "Agree Strongly" with a total scores range of 10 to 50. A higher score represents greater participant satisfaction.
Participant Satisfaction Score on GTS Survey 2 | Up to 130 days from baseline
  Assessed by the Genetic Testing Satisfaction (GTS) 2, a 10-item measure rated on a 5-point scale from 1 "Strongly Disagree" to 5 "Agree Strongly" with a total scores range of 10 to 50. A higher score represents greater participant satisfaction.
Multidimensional Impact of Cancer Risk Assessment (MICRA) Score | Up to 130 days from baseline
  Assessed by the Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire to measure the psychological impact of testing over the past week, and comprised of 25 question which are rated on a 4-point scale from 1 "Never" to 4 "Often" with a total scores range of 25 to 100. A higher score represents greater psychological impact.
Participant Decisional Regret Score | Up to 130 days from baseline
  Assessed by the Decisional Regret Survey to measure the degree of participant regret in choosing to undergo germline genetic testing, and comprised of 5 questions rated on a 5-point scale from 1 "Strongly Agree" to 5 "Strongly Disagree" with a total scores range of 5 to 25. A higher score represents greater regret.
Detection Rate of Germline Predisposition | Up to 63 months
  Defined as the number of participants with an identified germline predisposition on genetic testing who would not have met National Comprehensive Cancer Network (NCCN) guideline-based germline genetic testing recommendations.
Impact of Genetic Results on Clinical Decision-Making | Up to 130 days from baseline
  Assessed by the Primary Clinician Survey, a 5-question survey including 4 questions with graded answers (Strongly Agree, Agree, Neither, Disagree, Strongly Disagree) and 1 free text question for overall study feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Reilly, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu